CLINICAL TRIAL: NCT01426529
Title: Caveolin-1 and Vascular Dysfunction
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Luminita Pojoga, Instructor of Medicine, Associate Physiologist, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2010P002187; 1R01HL104032-01 (NIH)
Record Dates: First submitted 2011-08-30; First posted 2011-08-31 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Insulin Resistance
MeSH Terms: conditions — Hypertension; Insulin Resistance | interventions — p-Aminohippuric Acid; Angiotensin II; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- major allele homozygous (Experimental): we will compare this arm with the minor allele carrier arm
  Interventions: Drug: Para-aminohippuric Acid; Drug: Angiotensin II; Drug: Norepinephrine
- minor allele carriers (Experimental): we will compare this arm with the major allele homozygous arm
  Interventions: Drug: Para-aminohippuric Acid; Drug: Angiotensin II; Drug: Norepinephrine

INTERVENTIONS:
Drug: Para-aminohippuric Acid — Aminohippurate sodium is an agent to measure effective renal plasma flow (ERPF). It is the sodium salt of para-aminohippuric acid, commonly abbreviated "PAH".
  Other Names: PAH
Drug: Angiotensin II — Angiotensin II (Ang II) is a naturally occurring hormone whose primary purpose is to regulate the body's internal volume. It accomplishes this task by influencing the function of a variety of organs and tissues. It increases aldosterone secretion from the adrenal gland. It causes blood vessels to contract, particularly renal blood vessels, and it modifies the way the heart works.
  Other Names: AngII; AII
Drug: Norepinephrine — A hormone that is normally present in your body, which regulates your blood pressure.
  Other Names: NE

SUMMARY:
Caveolin-1 and Vascular Dysfunction

Thank you for your interest in the investigators Blood Pressure Research Study. The National Institutes of Health are sponsoring us to investigate why patients develop high blood pressure, atherosclerosis (hardening of the arteries), and heart disease. There are two parts of the investigators research program. The first part is a screening visit. At this visit you will be given a brief physical exam and will be asked questions concerning your medical history. During the same visit you will have your blood drawn for routine screening and genetic testing. You will also be asked to collect a urine sample for routine screening.

If the doctor finds that you are a healthy candidate you will be invited to participate in the second part of the study. During Phase II, the investigators will perform physiological tests after you are placed on a low salt diet and again after you are placed on a higher salt diet. If you are on blood pressure medication, it may be necessary to discontinue taking your present medication for up to three months before beginning the study. Patients discontinuing their current blood pressure medication may be placed on a different blood pressure medication during this 'washout' period if necessary to maintain blood pressure at pre-study levels.

Once your blood pressure medications are discontinued, you will be closely monitored. If you do not own a home blood pressure monitor, the investigators will provide one for you to use during the study so that you can keep a daily record of your blood pressure readings. The investigators will ask you to call us every three days to report your blood pressure readings. After you have stopped taking your medication, dieticians at the hospital will make you low salt meals to eat at home for about seven days. On the last day of the low salt diet, you will be asked to begin a 24-hour urine collection that you will bring with you when you are admitted to the hospital that evening. That morning, you will be required to come to the Center for Clinical Investigations (CCI) at Brigham and Women's Hospital for a one-hour test to check if your body is in the correct salt balance.

You will return that evening to the CCI where you will be admitted for your study that will occur the next morning. On the morning of your low salt study, the investigators will collect some blood samples. The investigators will also take ultrasound pictures of your heart to see how salt and hormones affect the way your heart and blood vessels functions. These tests will last approximately 5 hours and you will be discharged around 2:00 PM. For the next 5-7 days, you will be placed on a high salt diet. During this diet period, you will eat all your own food, but the investigators will give you some supplements to add to your meals. After 5-7 days on your high salt diet, on the morning of your second admission to the hospital, you will be asked to begin a final 24-hour urine collection. That morning, you will again be required to come to the CCI for a blood test, and you will return later that evening to the inpatient CCI where you will be admitted for your final overnight study. The same study that was done for the low salt diet will be repeated for the high salt study. You will be discharged at around 2:00 p.m. These studies will help to determine if you are salt-sensitive. In addition, the investigators hope to learn more about the hormones that regulate your blood pressure and the genes responsible for regulating those hormones.

You will have the option to spend a second night in the CCI after each diet phase in order to participate in an optional study of the blood vessels in the arm. This study also uses an ultrasound machine. It will last about 2 hours in the morning.

You will be placed back on your initial blood pressure medication (if you are on any) and returned to your regular physician for care. The investigators can also provide clinically relevant information to you.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* mild to moderate hypertension
* no other major illnesses
* BMI < or equal to 40

Exclusion Criteria:

* secondary illnesses
* BMI > 40
* taking 4 or more anti-hypertensive medications
* BP >160/100 on screening exam
* Alcohol intake >12 oz per week
* Current smoking
* Recreational drug use
* use of birth control pills or contraceptive hormone shots

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-10-01 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Genetic Variation at the Caveolin-1 Locus | 5 years
  We are testing our hypothesis that genetic variation at the cav-1 locus is a determinant of vascular phenotypes in hypertensive subjects. We will recruit hypertensive subjects who will be classified into two groups according to genotype status at rs926198 of CAV-1. Vascular function status will be determined using four markers: renal blood flow (primary endpoint), brachial artery reactivity, aortic compliance, and blood pressure levels.
  We will assess these endpoints before and after two provocations: low vs. high salt intake and AngII infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Luminita Pojoga, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Brown JM, Williams JS, Luther JM, Garg R, Garza AE, Pojoga LH, Ruan DT, Williams GH, Adler GK, Vaidya A. Human interventions to characterize novel relationships between the renin-angiotensin-aldosterone system and parathyroid hormone. Hypertension. 2014 Feb;63(2):273-80. doi: 10.1161/HYPERTENSIONAHA.113.01910. Epub 2013 Nov 4. PMID 24191286